CLINICAL TRIAL: NCT04449263
Title: Comparing the Performance of 1 Day Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-109
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Lens A (Test) (Experimental): Subjects will be randomized to wear Lens A (test) the control Lens B for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Interventions: Device: Lens A; Device: Lens B; Device: Habitual Lenses
- Lens B (Control) (Active Comparator): Subjects will be randomized to wear Lens B (control) and Lens A (Test) for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Interventions: Device: Lens A; Device: Lens B; Device: Habitual Lenses
- Habitual Lenses (Active Comparator): All subjects will wear their habitual lenses for two weeks prior to randomization of Test lens A and control lens B.
  Interventions: Device: Habitual Lenses

INTERVENTIONS:
Device: Lens A — Subjects will be randomized to wear Lens A (test) for 2 weeks.
  Other Names: FDA Approved, non-marketed, daily disposable multifocal lens
  Arms: Lens A (Test); Lens B (Control)
Device: Lens B — Subjects will be randomized to wear Lens B (control) for 2 weeks.
  Other Names: FDA Approved, daily disposable multifocal lens
  Arms: Lens A (Test); Lens B (Control)
Device: Habitual Lenses — All Subjects will wear their habitual lenses for 2 weeks prior to randomization of test lens and control lens.

SUMMARY:
The objective of the study was to compare the lens handling and performance of Lens A to habitually worn multifocal contact lenses and to the competitor Lens B.

DETAILED DESCRIPTION:
The objective of the study was to compare the lens handling and performance of Lens A to habitually worn multifocal contact lenses and to the competitor Lens B. This was a prospective, randomized, participant-masked, crossover, bilateral dispensing study conducted at up to 5 clinical practice sites in the United States. Subjects were dispensed their habitual lenses for two weeks prior to randomization of Test Lens and Control Lens. Each lens type will be worn for 2 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 42 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears multifocal soft contact lenses, for the past 3 months minimum;
7. Has refractive astigmatism no higher than -0.75DC;
8. Is presbyopic and requires a reading addition of at least +0.75D and no more than +2.50D;
9. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deem to be 'acceptable', with the available study lens parameters (sphere +4 to -6; near addition or LOW, MEDIUM, HIGH).

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Habitually wears one of the study contact lenses;
3. Has any known active* ocular disease and/or infection that contraindicates contact lens wear;
4. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
5. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
6. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
7. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
8. Has undergone refractive error surgery or intraocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Golden, Principal Investigator — Golden Vision; Keith Wan, Principal Investigator — Scripps Poway Eyecare; Shane Kannarr, Principal Investigator — Kannarr Eye Care; David Ardaya, Principal Investigator — Golden Optometric Group; Katherine Bickle, Principal Investigator — ProCare Vision Center
Locations (5):
- United States (5):
  - Scripps Poway Eyecare, San Diego, California
  - Golden Optometric Group, Whittier, California
  - Golden Vision, Sarasota, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - ProCare Vision Center, Granville, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 subjects were enrolled and 1 subject discontinued because of screen failure prior to dispense of their habitual lenses.
Pre-assignment Details: All 59 subjects wore their habitual lenses for two weeks prior to randomization to test lens and control lens.
Groups:
- Lens A (Test) Then Lens B (Control): Subjects wore their habitual lenses for 2 weeks and were randomized to wear Lens A (test) then Lens B (control) for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Contact lens: Habitual Lenses Contact Lens: Test Lens A Contact Lens: Control Lens B
- Lens B (Control) Then Lens A (Test): All Subjects wore their habitual lenses for 2 weeks prior to randomization and were randomized to wear Lens B (control) then Lens A (test) for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Contact Lens: Habitual lenses
  Contact lens: Control Lens B
  Contact Lens : Test lens A
Period: First Intervention
Arm/Group | Lens A (Test) Then Lens B (Control) | Lens B (Control) Then Lens A (Test)
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lens A (Test) Then Lens B (Control) | Lens B (Control) Then Lens A (Test)
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | Lens A (Test) Then Lens B (Control) | Lens B (Control) Then Lens A (Test)
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects wore their habitual lenses for two weeks and then randomized to wear Test lens A and Control Lens B for 2 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Subjective At-home Ratings for Ease of Lens Handling for Insertion
Description: Subjective at-home ratings for ease of Lens handling for insertion will be assessed using a 0-10 scale, (0=very difficult, 10=very easy)
Time Frame: Day 13
Population: One subject was not included in the analysis for all study arms because of protocol deviation. One more subject was excluded form the analysis from Len B control Arm only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjects Habitual Lenses: Subjects will wear their habitual lenses for 2 weeks prior to randomization of test lens and control lens.
  Contact Lenses: Habitual Lenses
- Lens A (Test): Subjects were randomized to wear Lens A (test) then Lens B (control) for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Contact Lens: Test Lens A
- Lens B (Control): Subjects were randomized to wear Lens B (control) then Lens A (test) for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Contact lens: Control Lens B
Arm/Group | Subjects Habitual Lenses | Lens A (Test) | Lens B (Control)
Number analyzed (Participants) | 58 | 58 | 57
units on a scale | 8.90 (1.59) | 8.28 (2.10) | 9.18 (1.12)

ADVERSE EVENTS:
Time Frame: All subjects wore their habitual lenses for two weeks and then randomized to wear test lens A and control lens B for 2 weeks, a total of 6 weeks.
Groups:
- Subjects Habitual Lenses: All Subjects wore their habitual lenses for 2 weeks prior to randomization of test lens and control lens.
  Contact Lenses: Habitual Lenses
Arm/Group | Subjects Habitual Lenses | Lens A (Test) | Lens B (Control)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04449263/Prot_SAP_000.pdf